CLINICAL TRIAL: NCT02655718
Title: Short and Long Term Outcomes of Acute Coronary Syndrome in Patients With Non Obstructive Coronary Atherosclerosis
Acronym: NOCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Vyacheslav Ryabov, MD, PhD Research Institute for Cardiology, Russian Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2411
Record Dates: First submitted 2015-12-29; First posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Acute Coronary Syndrome
Keywords: ACS; Non obstructive coronary atherosclerosis
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with ACS (Other): Patients with ACS who underwent coronary angiography within 72 hours from the onset of disease. In identifying nonobstructive coronary atherosclerosis , patients underwent cardiac contrast MRI.
  Interventions: Other: Patients with ACS; Device: MRI

INTERVENTIONS:
Other: Patients with ACS — Cardiovascular magnetic resonance (CMR) imaging with contrast (Gadovist) in regime inversion recovery time, regime T-2 weighted images , T1-weighted images.
Device: MRI

SUMMARY:
The purpose of the study is to assess short and long term outcomes of acute coronary syndrome in patients with non obstructive coronary atherosclerosis, to optimize the algorithm for diagnosis and to evaluate its effectiveness

DETAILED DESCRIPTION:
The study non randomized, opened, controlled. Cardiovascular Magnetic - resonance imaging reveals both ischemic and non-ischemic causes of acute coronary syndrome. Currently, it is the best method for Imaging and damage assessment of myocardial viability in coronary atherosclerosis and noncoronary injuries (V.Yu.Usov 2012).

Taking into account the results of previous (D. Kawecki, B. Morawiec, P. Monney, 2015) research, it can be concluded that the introduction of cardiovascular magnetic resonance imaging into routine practice will change the structure of morbidity among patients with acute coronary syndrome and non obstructive coronary atherosclerosis . The research was conducted on small groups of patients, and therefore further data acquisition is required.

It is planned to study 200 patients with acute coronary syndrome. On admission, they will receive the standard treatment of ACS with and without ST elevation. Within 72 hours they will performed diagnostic coronary angiography. If in case of non stenotic atherosclerosis of coronary artery (normal / stenosis < 50%) patients are planned for cardiac contrast MRI, which will identify both ischemic and non-ischemic causes of acute coronary syndrome. At 30 days, 6 months, 12 months the researchers will assess the clinical condition of the patients, perform cardiac ultrasound for the evaluation of myocardial contractile function, evaluate the incidence rate of secondary endpoints

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years at time of randomization (18 years and older)
* acute coronary syndrome
* no obstructive coronary atherosclerosis (normal coronary artety/ plaques <50%) is based on the results of coronary angiography for 3 days of admission
* written the informed consent to participate in research

Exclusion Criteria:

* patients previously undergone endovascular / surgical revascularization of coronary artery
* severe comorbidity
* Contacts/Locations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of inflammatory infiltrate, ischemia, infarction in the myocardial tissue | 14 days after ACS
Left ventricular ejection fraction (Echo) | 14 days after ACS

SECONDARY OUTCOMES:
Incidence of the acute myocardial infarction | 14 days after ACS
Incidence of unstable angina | 14 days after ACS
Incidence of Takotsubo syndrome | 14 days after ACS
Incidence of myocarditis | 14 days after ACS
Incidence of the mortality | 6 month and 12 month after ACS
Incidence of the recurrent myocardial infarction | 6 month and 12 month after ACS
Incidence of the heart failure | 6 month and 12 month after ACS
Incidence of the stroke | 6 month and 12 month after ACS

CONTACTS AND LOCATIONS:
Overall Officials: Vyacheslav Ryabov, MD,PhD, Principal Investigator — Research Institute for Cardiology
Locations (1):
- Research Institutite for Cardiology, Tomsk, Tomskii Region, Russia